CLINICAL TRIAL: NCT05277532
Title: Elucidating the Interplay Between Circadian Rhythm and Physical Exercise on Metabolism in Patients With Type 1 Diabetes and Overweight
Brief Title: Effect of Circadian Rhythm and Physical Exercise in Overweight Type 1 Diabetes Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Toft, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2021-05137
Record Dates: First submitted 2022-02-18; First posted 2022-03-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes; Overweight
Keywords: high intensity interval training; metabolomics
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: A randomized crossover design (comparing morning vs afternoon exercise) in parallel groups (Type 1 diabetes and control subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 1 diabetes with overweight (Active Comparator): High intensity interval training (HIIT), a single bout, randomly performed either in the morning or in the afternoon in a cross-over design.
  Interventions: Behavioral: High intensity interval training (HIIT)
- Overweight but otherwise healthy control subjects (Active Comparator): High intensity interval training (HIIT), a single bout, randomly performed either in the morning or in the afternoon in a cross-over design.
  Interventions: Behavioral: High intensity interval training (HIIT)

INTERVENTIONS:
Behavioral: High intensity interval training (HIIT) — HIIT performed either in the morning or in the afternoon

SUMMARY:
Cardiometabolic risk in patients with abdominal obesity and type 1 diabetes can be moderated by life style modifications. There is an intimate link between gene regulation and circadian rhythm in mediating response to exercise in a variety of insulin sensitive organs.

The aim of this project is to evaluate, by intervention, the interplay of circadian rhythm and high intensity interval training (HIIT) on glucose control and skeletal muscle metabolism in patients with overweight with or without type 1 diabetes (T1D).

DETAILED DESCRIPTION:
High intensity interval training (HIIT) is a promising intervention for lifestyle treatment in type 1 diabetes. In spite of the interplay between circadian rhythms and exercise, the time of day in which the most robust adaption to HIIT can be achieved is unknown. The main goal of the study is to compare the efficacy of morning and afternoon HIIT in regulating blood glucose values in participants with type 1 diabetes and overweigt and to compare the effect in overweight but otherwise healthy subjects. Additionally, the investigators aim to to elucidate the metabolomics in the different settings. Healthy controls will be used to compare whether the effect of HIIT and interplay with circadian rhythm on organ metabolism is impaired in patients with T1D.

A randomized cross-over trial with 25 participants with type 1 diabetes and 25 control subjects will be performed. The participants will be examined on three occasions on an out-patient basis . Visit 1 aim to run baseline measurements and a bicycle test to define maximum exertion . On visit 2 the participants will perform a single bout of HIIT (6 1-minute pulses at maximal exertion, interspersed with 1-minute recovery) either in the morning (09.00) or afternoon (16.00). After a 1-week washout period, the participants will return for visit 3 and an opposing exercise time. Primarily, the efficacy of the morning and afternoon HIIT will be judged by the continuous glucose monitor (CGM) -based glycaemia measurements. Additionally, during the visits the investigators will collect repeated blood samples to assess the effect of exercise timing on the diurnal hormonal rhythms. Muscle biopsies will be collected before and directly after HIIT.

The hypothesis is that afternoon HIIT will be more efficacious in controlling blood glucose based on the preliminary data gathered from a 'free living' pilot study in type 2 diabetes. The current study will aim to compare the morning and afternoon exercise in controlled conditions, eliminating the effects of dietary intake, medication and sleep cycle disruption. Additionally, the tissue factors responsible for the differing glycaemic response to morning and afternoon exercise will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-30
* type 1 diabetes or healthy subjects

Exclusion Criteria:

* nicotine usage,
* cardiovascular disease (CVD),
* blood pressure >160/95,
* pregnancy,
* treatment with other pharmaceutical drugs than insulin, stable dose of thyroid hormone, statins, and antihypertensive drugs (excluding beta blockers).

Additional exclusion criteria for diabetes subjects:

* diabetes duration less than 6 months,
* proliferative or severe non-proliferative retinopathy,
* chronic kidney disease with glomerular filtration rate (GFR) <60 ml/min,

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Time in Glucose target range (4-10 mmol/L) for tissue glucose from CGM. | 48 hours
  Time in target glucose range (expressed as % of total time) measured by continuous subcutaneous glucose sensors following morning or afternoon HIIT respectively. Measurements are uploaded from the CGM device and analyzed.

SECONDARY OUTCOMES:
Tissue specific effects of HIIT in type 1 diabetes vs healthy subjects | 2 hours; muscle and blood samples are collected directly before and after HIIT, respectively.
  Plasma and skeletal muscle samples will be subjected to transcriptomic and/or metabolomic analyses to evaluate the impact of HIIT on metabolic outcomes.
Time below Glucose target range (< 4 mmol/L) for tissue glucose from CGM. | 48 hours
  Time in the hypoglycaemic range (expressed as % of total time) measured by continuous subcutaneous glucose sensors following morning or afternoon HIIT respectively. Measurements are uploaded from the CGM device and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Dahlman, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta sjukhus, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No